CLINICAL TRIAL: NCT04501562
Title: TO-ChERIsH: Trajectory of Cardiovascular Ageing, Its Determinants and Impact on Health
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2252
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Ageing
Keywords: Echocardiogram; MRI/MRS
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subject
  Interventions: Other: Examinations; Other: Cardiovascular Tests; Other: Bio-specimen collection; Other: Clinical/health outcome collection

INTERVENTIONS:
Other: Examinations — Participants will undergo focused examinations that include measurement of height, weight, waist circumference, body composition analysis, baseline data collection and blood pressure examinations. Resting electrocardiography will be performed to ascertain sinus rhythm.
Other: Cardiovascular Tests — Specific quantitative cardiac ageing-related outcome parameters will be examined by multimodal techniques including two-dimensional transthoracic echocardiogram, and/or non-contrast magnetic resonance imaging/magnetic resonance spectroscopy.
Other: Bio-specimen collection — Bio-specimens collected will include fresh blood, urine and/or stool specimens.
Other: Clinical/health outcome collection — Health status will be tracked by telephone follow-up and/or matching at national disease registries at periodic intervals within one to five years, up to three decades.

SUMMARY:
Specific Aim 1: To determine longitudinal changes in CV ageing (changes in CV imaging) over time.

Hypothesis: There are differences in rates of CV ageing over time.

Specific Aim 2: To study determinants of CV ageing To assess how biological pathways affect CV ageing by studying the relationships between biological signatures measured in longitudinal biospecimens are associated with CV ageing.

Hypothesis: Antecedent biological markers are associated with progression of CV ageing.

Specific Aim 3: To determine the impact of CV ageing progression on the development of clinical CVD and the overall physical, cognitive and functional health of the elderly.

Hypothesis: Those with stable CV imaging phenotypes have lower incidence of clinical CVD and also better overall health in ageing, compared to those with rapid deterioration (unhealthy CV ageing).

DETAILED DESCRIPTION:
In Singapore, elderly residents aged 65 years and above make up 10.5% of our population and this is expected to double in 2030 (Singapore Department of Statistics, Ministry of Manpower, Registry of Birth and Deaths, September 2014). Cardiovascular diseases account for the majority of disability-adjusted life years by broad cause group, accounting for 20% of 399,675 life years lost due to mortality and ill-health in 2010 (Source: Estimates from the Singapore Burden of Disease Study 2010).

While chronological ageing is inevitable, a clear understanding is needed as to how ageing becomes a critical risk component of CVD for some individuals, and the mechanisms through which ageing results in such a vulnerable phenotype that leads towards clinical CVD. Following that, clinical tools and clinical guidelines to reduce cardiovascular disease and other health burdens contributed by ageing may be formulated. Such strategies may potentially reduce burdens and cost of healthcare provision to the ageing population.

Our proposal will generate data that identifies functional and structural changes in the cardiovascular system that occur in during ageing. Using a longitudinal design, this research will provide high quality evidence that distinguishes healthy from unhealthy cardiovascular ageing, and reveal determinants and impact of CV ageing over time on CVD and associated health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >= 21 years old

Exclusion Criteria:

* Unable to provide written informed consent to participate in the study

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited through population based studies (Singhealth IRB 2018/3173).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2049-12 (Estimated); Study Completion 2049-12 (Estimated)

PRIMARY OUTCOMES:
To identifies functional and structural changes in the cardiovascular system that occur in during ageing. | 5 Years
  Health status will be tracked by telephone follow-up and/or matching at national disease registries at periodic intervals within one to five years, up to three decades.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Koh, M.D., Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No